CLINICAL TRIAL: NCT05080387
Title: Neopterin in Acute Coronary Syndrome Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina Khairy Alyshaa Gorgy, Mina Khairy Alyshaa Gorgy, Assiut University
Other Study IDs: Neopterin
Record Dates: First submitted 2021-10-05; First posted 2021-10-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2021-10

CONDITIONS: Neopterin in Acute Coronary Syndrome Patients
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood sample — Blood samples will obtained for measurement of neopterin level through ELIZA

SUMMARY:
Measurement of neopterin in ACS patients

DETAILED DESCRIPTION:
1. Detect level of neopterin in ACS patients to detect whether there is relation or not between ACS and neopterin
2. Detection of relation between neopterin and cardiac enzymes as CK and troponine in ACS patients
3. Detect relation between neopterin level and in hospital events

ELIGIBILITY:
Inclusion Criteria:

* All patient of sample size admitted to cardiology departmentof Assiut university hospital with :

  1. Acute typical chest pain
  2. Positive cardiac enzymes
  3. ECG show recent ischemic changes
  4. ECHO show SWMA

Exclusion Criteria:

1. Patients not fulfill inclusion criteria.
2. Patients with other diseases which may cause increase of neopterin level as viral infections, intracellular bacteria or parasites infections, certain malignancies, allograft rejection

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients of sample size admitted to cardiology department with ACS.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
To detect whether there is association between neopterin and ACS or not | 72 hours
  To detect whether there is association between neopterin and ACS or not

SECONDARY OUTCOMES:
Detection of relation between neopterin and cardiac enzymes as CK and troponine in ACS and detection of relation between neopterin level and in hospital events | 72 hours
  Detection of relation between neopterin and cardiac enzymes as CK and troponine in ACS and detection of relation between neopterin level and in hospital events

CONTACTS AND LOCATIONS:
Overall Officials: Magdy Ibrahim Aldesowky, Lecturer, Principal Investigator — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Share if participants agree